CLINICAL TRIAL: NCT04542018
Title: Effects of Low FODMAP Diet on Colonic Epithelial Physiology in Diarrhea-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Prashant Singh, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00166423; K23DK129327 (NIH)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Patients with diarrhea predominant IBS (IBS-D) will undergo 4 weeks of low FODMAP diet. Urine, blood, stool, and colon biopsies will be collected before and after the diet to assess changes in gut physiology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study patients with IBS-D (Experimental): Patients with diarrhea-predominant IBS who will undergo a low FODMAP diet for 4 weeks
  Interventions: Other: a low FODMAP diet for 4 weeks

INTERVENTIONS:
Other: a low FODMAP diet for 4 weeks — low FODMAP diet for 4 weeks

SUMMARY:
This research is studying whether changing an individual's diet may have an impact as a treatment or outcome for Irritable Bowel Syndrome (IBS). This research will show if diet might play a role in triggering changes that may cause IBS. This study is being done to learn if a low FODMAP (fermentable, oligosaccharides, disaccharides, monosaccharides, and polyols) diet causes changes in the colon lining which mediates improvement in IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Normal serum studies including serum tissue-transglutaminase antibodies, thyroid stimulating hormone levels, C-reactive protein or fecal calprotectin, complete blood count since the onset of symptoms.
* Normal stool studies including, ova and parasites since the onset of symptoms
* IBS-SSS score of ≥175 at the end of the 7-day screening period

In case of presence of any alarm features and/or elevated inflammatory markers (C-reactive protein or fecal calprotectin), patients will be eligible if they have been excluded for inflammatory bowel disease with colonoscopy in the last one year.

Exclusion criteria

* individuals already on a LFD or other dietary restriction such as gluten free diet within the past 6 months
* individuals with any known food allergy or insulin-dependent diabetes
* known history of celiac disease, inflammatory bowel disease or microscopic colitis
* prior small bowel or colonic surgery or cholecystectomy
* pregnant patients
* Antibiotics in the past 3 months
* Those who regularly use mast cell stabilizers or anti-histaminic or non-steroidal anti-inflammatory agents (NSAIDs) excluding daily baby aspirin or steroids or bile-acid binder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Singh, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao J, Lee AA, Abtahi S, Turner JR, Grover M, Schmidt A, Schmidt TM, Nee JW, Iturrino J, Lembo A, Chey WD, Wiley JW, Singh P. Low Fermentable Oligosaccharides, Disaccharides, Monosaccharides, and Polyols Diet Improves Colonic Barrier Function and Mast Cell Activation in Patients With Diarrhea-Predominant Irritable Bowel Syndrome: A Mechanistic Trial. Gastroenterology. 2026 Jan;170(1):132-147. doi: 10.1053/j.gastro.2025.07.016. Epub 2025 Jul 30. PMID 40749856

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants began the same 4-week Low FODMAP diet treatment. Once participants completed the 4-week intervention, they were categorized based on the changes in their IBSSS survey responses. Data was analyzed for each group separately. Participants who did not submit their IBSSS surveys after 4-weeks of treatment could not be placed in either group, submitted no data, and are not considered to have "completed" the trial.
Groups:
- Responders: Patients with diarrhea-predominant IBS who will undergo a low FODMAP diet for 4 weeks
  a low FODMAP diet for 4 weeks: low FODMAP diet for 4 weeks
  Participants in this arm reported a change in IBS-SSS score between the baseline survey and the survey after 4 weeks of following the Low FODMAP diet of at least 100 points.
- Non-Responders: Patients with diarrhea-predominant IBS who will undergo a low FODMAP diet for 4 weeks
  a low FODMAP diet for 4 weeks: low FODMAP diet for 4 weeks
  Participants in this arm reported a change in IBS-SSS score between the baseline survey and the survey after 4 weeks of following the Low FODMAP diet of less-than 100 points.
- Intervention Recipients Who Did Not Complete the Trial: These participants began the 4 week Low FODMAP diet treatment, but did not complete the treatment or report data to study team. They were, therefore, not categorized into "responders" or "non-responders".
Period: Overall Study
Arm/Group | Responders | Non-Responders | Intervention Recipients Who Did Not Complete the Trial
Started | 34 | 8 | 6
Completed | 34 | 8 | 0
Not Completed | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Responders | Non-Responders | Intervention Recipients Who Did Not Complete the Trial | Total
Number analyzed (Participants) | 34 | 8 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11.2) | 44.6 (11.8) | 32.2 (10.3) | 38.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 4 | 35
  Male | 11 | 0 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 32 | 8 | 6 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 2 | 6
  White | 24 | 8 | 3 | 35
  More than one race | 3 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 8 | 6 | 48
Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) [Mean (Standard Deviation); unit: score on a scale] — IBS-SSS is a scale for assessing overall IBS symptom severity. It includes 5 questions concerning symptoms over the past 10 days: average severity of abdominal pain, # of days with abdominal pain, average severity of abdominal distension or bloating, satisfaction with bowel habits, and the overall interference in their quality of life from these symptoms. Questions are scored on a 0-100 scale and are summed to a total score between 0-500. Lower scores indicate lower symptom severity.
  Participants were separated into arms based on the change in their responses from baseline to 4 weeks. Population: Because 6 participants who did not finish the trial did not provide week 4 IBS-SSS, they are not included in the analysis
  score on a scale | 334.2 (81.36) | 254.5 (65.52) | 303.6 (113.1) | 317.4 (86.2)

OUTCOME MEASURES:

1. Primary Outcome: Lactulose Mannitol Excretion
Description: Changes in cumulative excretion of lactulose and mannitol in timed urine collection before and after low FODMAP diet measured during 8-24h
Time Frame: 4 weeks
Population: No data was collected from "Intervention Recipients Who Did Not Complete The Trial" arm
Measure: Median (Full Range); unit: micrograms per ml
Groups:
- Responders: Patients with diarrhea-predominant IBS who will undergo a low FODMAP diet for 4 weeks
  Participants in this arm reported a change in IBS-SSS score between the baseline survey and the survey after 4 weeks of following the Low FODMAP diet of at least 100 points.
- Non-Responders: Patients with diarrhea-predominant IBS who will undergo a low FODMAP diet for 4 weeks
  Participants in this arm reported a change in IBS-SSS score between the baseline survey and the survey after 4 weeks of following the Low FODMAP diet of less-than 100 points.
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 34 | 8
micrograms per ml
  Baseline - Lactulose Excretion: number analyzed (Participants) | 28 | 6
  Baseline - Lactulose Excretion | 512.5 [99 to 3456] | 394.5 [204 to 1982]
  4-Week - Lactulose Excretion: number analyzed (Participants) | 28 | 6
  4-Week - Lactulose Excretion | 456.8 [60 to 1568] | 411 [221.4 to 992.5]
  Baseline - Mannitol Excretion: number analyzed (Participants) | 28 | 6
  Baseline - Mannitol Excretion | 41395 [9600 to 430100] | 86820 [79040 to 207900]
  4-Week - Mannitol Excretion: number analyzed (Participants) | 28 | 6
  4-Week - Mannitol Excretion | 37030 [2704 to 83356] | 54825 [11314 to 500480]

2. Secondary Outcome: Changes in Epithelial Permeability - Tight Junction Gene Expression
Description: Changes in tight junction (TJ) gene expression in colonic biopsies before and after low FODMAP diet Gene expression of Tight junction proteins were normalized to that of Glyceraldehyde 3-phosphate dehydrogenase (GAPDH).
Time Frame: 4 weeks
Population: No data was analyzed for the "Intervention Recipients Who Did Not Complete The Trial" arm because those participants did not submit second sample.
Measure: Median (Full Range); unit: ratio of TJ proteins to GAPDH
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 34 | 8
ratio of TJ proteins to GAPDH
  Baseline - ZO-1 | .9 [.1 to 3.5] | .7 [.1 to 1]
  4-week - ZO-1 | 1.4 [.3 to 4.8] | 1.1 [.2 to 3.2]
  Baseline - JAM-A: number analyzed (Participants) | 32 | 8
  Baseline - JAM-A | 0.9 [0.03 to 2.6] | 0.5 [0.1 to 1.3]
  4-week - JAM-A: number analyzed (Participants) | 32 | 8
  4-week - JAM-A | 2 [0.2 to 7.2] | 1.3 [0.1 to 3.3]
  Baseline - Occludin | 0.9 [0.1 to 3] | 0.6 [0.1 to 1.1]
  4-week - Occludin | 1.3 [0.1 to 4.8] | 0.8 [0.1 to 2.1]
  Baseline - Claudin-1 | 0.6 [0.01 to 3.8] | 0.5 [0.1 to 3.7]
  4-week - Claudin-1 | 1.1 [0.04 to 3.7] | 0.9 [0.1 to 2.5]

3. Secondary Outcome: Changes in Epithelial Permeability - Quantitative Tight Junction Immunostaining
Description: Changes in Quantitative tight junction immunostaining of tight junctions in colonic biopsies before and after low FODMAP diet
  Data is reported as ratio of TJ proteins to NA-K ATPase.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio of TJ proteins to NA-K ATPase
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 34 | 8
ratio of TJ proteins to NA-K ATPase
  Baseline - ZO-1: number analyzed (Participants) | 22 | 4
  Baseline - ZO-1 | 0.06579 [0.008542 to 0.3880] | 0.03703 [0.01876 to 0.07138]
  4-week - ZO-1: number analyzed (Participants) | 22 | 4
  4-week - ZO-1 | 0.07330 [0.01938 to 0.3061] | 0.05063 [0.04520 to 0.07585]
  Baseline - JAM-A: number analyzed (Participants) | 22 | 4
  Baseline - JAM-A | 0.07493 [0.01628 to 0.2034] | 0.08437 [0.02690 to 0.09409]
  4-week - JAM-A: number analyzed (Participants) | 22 | 4
  4-week - JAM-A | 0.09149 [0.02220 to 0.3186] | 0.07267 [0.05500 to 0.09367]
  Baseline - Occludin: number analyzed (Participants) | 23 | 4
  Baseline - Occludin | 2.623 [0.6874 to 16.95] | 3.834 [2.624 to 9.378]
  4-week - Occludin: number analyzed (Participants) | 23 | 4
  4-week - Occludin | 5.529 [0.7352 to 13.05] | 5.533 [2.724 to 16.5]
  Baseline - Claudin-1: number analyzed (Participants) | 23 | 4
  Baseline - Claudin-1 | 6.542 [0.5603 to 20.69] | 10.40 [7.514 to 12.13]
  4-week - Claudin-1: number analyzed (Participants) | 23 | 4
  4-week - Claudin-1 | 11.22 [1.696 to 17.38] | 9.218 [1.108 to 20.86]

4. Secondary Outcome: Changes in Stool Microbiome - Alpha Diversity
Description: Changes in relative abundance of bacteria before and after low FODMAP diet. Alpha diversity was measured as number of Amplicon Sequence Variant (ASV) measured in the specimen.
Time Frame: 4 weeks
Population: No data was analyzed for the "Intervention Recipients Who Did Not Complete the Trial" arm because participants did not submit necessary samples for analysis.
Measure: Mean (Standard Deviation); unit: ASVs Observed
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 34 | 8
ASVs Observed
  Baseline - Alpha Diversity: number analyzed (Participants) | 23 | 4
  Baseline - Alpha Diversity | 649.087 (160.1794) | 532.75 (153.69)
  4-week - Alpha Diversity | 599.7391 (159.1749) | 608.5 (182.12)

5. Secondary Outcome: Changes in Stool Microbiome - Beta Diversity
Description: Changes in relative abundance of bacteria before and after low FODMAP diet. For the beta diversity, an analysis of similarities (ANOSIM)test based on Bray-Curtis distances is the best measure if the communities were different. The ANOSIM R statistic gives the scale of difference. ANOSIM R ranges from -1 to 1, where 1 means there is most interparticipant similarity within the group compared with between the different groups, and where -1 means there is least interparticipant similarity within the group compared with between the different groups. A value close to 0 indicates no significant difference between groups, meaning the dissimilarity is similar both within and between groups
Time Frame: 4 weeks
Population: No data was analyzed for the "Intervention Recipients Who Did Not Complete the Trial" arm because participants did not submit necessary samples for analysis.
  Some participants in both analyzed arms did not provide samples of sufficient quality for analysis.
Measure: Number; unit: units on a scale
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 23 | 4
units on a scale | -0.03722 | -0.2708

6. Secondary Outcome: Immunohistochemistry for Mast Cells
Description: Number of mast cells in sample after immunohistochemistry were counted.
Time Frame: 4 weeks
Population: No data was analyzed for "Intervention Recipients Who Did Not Complete the Trial", as they did not submit necessary samples.
Measure: Median (Full Range); unit: mast cell count per high power field
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 34 | 8
mast cell count per high power field
  Baseline - Mast Cell Count: number analyzed (Participants) | 23 | 5
  Baseline - Mast Cell Count | 23 [5.2 to 42.5] | 26.5 [18.7 to 27.2]
  4-Week - Mast Cell Count | 14.5 [5.4 to 25.8] | 11.5 [9.5 to 24.2]

7. Secondary Outcome: Gastrointestinal Patient Reported Outcomes Measurement Information System (PROMIS)
Description: PROMIS scales of Belly pain (5a) and diarrhea (6a) will be administered to assess the severity of belly pain and diarrhea in our patients. PROMIS Belly pain questionnaire and PROMIS diarrhea questionnaire have five and six questions, respectively, which assess symptom severity on a 5 point Likert scale. 50 indicates the general population mean with a standard deviation of 10. Higher T-scores on these questionnaires refer to more severe gastrointestinal symptoms.
  PROMIS belly pain asks how often did you have belly pain, severity of belly pain, interference with activities, bothersomeness and discomfort.
  PROMIS diarrhea asks how many days did you have loose stools, interference with activities, bothersomeness, and how often you experience urgency.
Time Frame: 4 weeks
Population: Participants in the "Intervention Recipients who did not Complete the Trial" arm did not submit surveys at the 4-week point.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Responders | Non-Responders | Intervention Recipients Who Did Not Complete the Trial
Number analyzed (Participants) | 34 | 8 | 6
T-score
  Baseline - Belly Pain | 63.6 (6.2) | 64.1 (5.1) | 63.7 (6.4)
  4-week - Belly Pain: number analyzed (Participants) | 34 | 8 | 0
  4-week - Belly Pain | 47.1 (9.4) | 60.8 (3.1) |
  Baseline - Diarrhea | 61.2 (10.8) | 49.1 (8.3) | 61.3 (5)
  4-week - Diarrhea | 55.8 (8.3) | 55.6 (8.4) | 0 (0)

8. Other Pre Specified Outcome: Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) - 4-Week
Description: Measure Description: IBS-SSS is a scale for assessing overall IBS symptom severity. It includes 5 questions concerning symptoms over the past 10 days: average severity of abdominal pain, # of days with abdominal pain, average severity of abdominal distension or bloating, satisfaction with bowel habits, and the overall interference in their quality of life from these symptoms. Questions are scored on a 0-100 scale and are summed to a total score between 0-500. Lower scores indicate lower symptom severity.
  Participants were separated into arms based on the change in their responses from baseline to 4 weeks.
Time Frame: 4 weeks
Population: Because 6 participants who did not finish the trial did not provide week 4 IBS-SSS, they were sorted into the third arm and not included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 34 | 8
score on a scale | 87.7 (84.8) | 235.4 (72.12)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Participants were encouraged to contact the study team if they experienced adverse events and were provided with contact information in the informed consent document. The study team did not specifically ask participants about adverse events or search medical records for potential AEs. Therefore, while all data collected is reported below, participants could have chosen not to report adverse events they experienced.
Arm/Group | Responders | Non-Responders | Intervention Recipients Who Did Not Complete the Trial
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 2/34 | 0/8 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Responders (N=34) | Non-Responders (N=8) | Intervention Recipients Who Did Not Complete the Trial (N=6)
Post-Vaccination Stomach Pain and Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT04542018/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT04542018/ICF_000.pdf